CLINICAL TRIAL: NCT03867643
Title: Efficacy of Hepatitis B Vaccine Boosters Among Neonatally Vaccinated Children in Chongqing
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qiu Li, Director, Children's Hospital of Chongqing Medical University
Other Study IDs: 2019-09
Record Dates: First submitted 2019-03-05; First posted 2019-03-08 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Hepatitis B Vaccine Adverse Reaction
Keywords: Hepatitis B Vaccine; booster; Immune response
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Separating serum, stored at -80 degrees Celsius
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hepatitis B vaccine booster: Children with anti-HBs at a level of<10mIU/mL or [10,100) mIU/mL before booster.
  Interventions: Biological: hepatitis B vaccine(HepB)
- Observation: Children with anti-HBs at a level of >100mIU/mL or [10,100) mIU/mL before booster.

INTERVENTIONS:
Biological: hepatitis B vaccine(HepB) — Children with anti-HBs at a low level (<10mIU/mL and [10,100) mIU/mL) were received a dose of hepatitis B vaccine booster after informed consent.
  Groups: Hepatitis B vaccine booster

SUMMARY:
Worldwide, hepatitis B virus (HBV) infection is a major cause of acute hepatitis, and chronic infection with HBV often leads to chronic hepatitis, liver cirrhosis, and hepatocellular carcinoma. So far, the most effective way to prevent HBV infection in susceptible population is to inject hepatitis B vaccine. However, long-term protection against hepatitis B virus (HBV) after vaccination remains widely debated. This study aims to carry out a comprehensive study to evaluate the efficacy of hepatitis B vaccine booster from the aspect of humoral and cellular immunity in neonatally vaccinated children in Chongqing.

DETAILED DESCRIPTION:
Hepatitis B virus (HBV) infection is a major public health problem around the world. More than 2 billion people have been infected with HBV. Although the World Health Organization (WHO) has incorporated hepatitis B vaccination into routine immunization programs for infants and adolescents since 1986 to reduce the incidence of chronic liver diseases, liver cirrhosis and hepatocellular carcinoma associated with hepatitis B virus, there are still more than 400 million chronic carriers. Although it is currently recognized that the most effective way to prevent HBV infection in susceptible population is to inject hepatitis B vaccine, the protective effect of the neonatally vaccinated children weakened as time goes on, which involves the question of the need of boosters. However, there are still some problems concerning hepatitis B vaccine boosters for healthy children. In China, there has not been a standardized directory to guide hepatitis B vaccine booster. Scholars have great controversy on the necessity, age, dosage and other aspects of hepatitis B vaccine booster. Researchers conducted an investigation on the Anti-HBs level of 93,326 Chinese children aged 1 - 16 who completed basic immunization. The results showed that the proportion of HBsAb positive in children aged 1 - 8 years old decreased dramatically, with 8 - year - old children having the lowest proportion of protective antibody. Therefore, this study is intended to explore the protective effect of hepatitis B vaccine on the body and the effect of multiple vaccines. This study will recruit some healthy children with anti-HBs at a low level (titer <10mIU/mL and [10,100) mIU/mL) in Chongqing and conduct selective re-vaccination according to the results of the first detection of hepatitis B surface markers in healthy children. According to the changes of immune status after booster, the efficacy of hepatitis B vaccine boosters was comprehensively evaluated.

ELIGIBILITY:
1. Born after Jan. 1st, 2005 in Chongqing, China;
2. Completion of the full primary immunization of HepB after birth;
3. No HBV booster vaccine history.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. History of allergy or adverse reaction of vaccine;
  2. History of immunosuppressive treatment or immunodeficiency;
  3. Any kind of vaccination in the past four weeks;
  4. Any acute disease or anti-infective therapy in the past four weeks;
  5. Fever history in the past one week (axillary temperature ≥ 38 ℃);
  6. Blood transfusion history;
  7. History of infectious diseases (hepatitis, AIDS, syphilis, gonorrhea, etc.);
  8. The family history of HBV in three generations of lineal relatives;
  9. Abnormal physical examination.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
HBsAb positive rate | 3-year
  The proportion of HBsAb in children with and without hepatitis B vaccine boosters
HBsAg-specific T cell response | 3-year
  The proportion of HBsAg-specific IFN-γ-producing T cells in children with and without hepatitis B vaccine boosters
HBsAb protective efficacy | 3-year
  Evaluate the changes in the protective efficacy of HBsAb after hepatitis B vaccine booster

CONTACTS AND LOCATIONS:
Overall Officials: Yao Zhao, postdoctor, Study Director — Chongqing Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China